CLINICAL TRIAL: NCT04877912
Title: Development and Testing of an Accurate, Rapid and Inexpensive MRI Protocol for Breast Cancer Screening - A Pilot Study
Brief Title: Accurate, Rapid and Inexpensive MRI Protocol for Breast Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB16-0396
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: MRI Screening; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Biopsy Group: We will scan 50 women who are scheduled for a breast biopsy. Subjects will receive an MRI exam that is research-only prior to the biopsy.
  Interventions: Diagnostic Test: MRI Abbreviated Scan
- MRI Unknown Cancer Status Group: We will scan 150 women with dense breasts and/or women who have intermediate risk of breast cancer for this study. Subjects will receive an MRI exam that is research-only.
  Interventions: Diagnostic Test: Abbreviated MRI Scan

INTERVENTIONS:
Diagnostic Test: MRI Abbreviated Scan — All subjects will be receiving an MRI scan, up to 15 minutes long that includes an injection of contrast agent. This contrast agent will be injected into the arm and will help the doctors to read the MRI more effectively. If there is a lesion (abnormality) in the breast, the contrast agent will go to the lesion first and we will be able to see it better.
  The examination table will then move subject into the magnet, which is a long tube with a diameter of about 3 feet. Subject will be asked to lie in the magnet for about 15 minutes. During the periods when we are taking pictures, we will ask subject to be as still as possible.
  Groups: Biopsy Group
Diagnostic Test: Abbreviated MRI Scan — All subjects will be receiving an MRI scan, up to 15 minutes long that includes an injection of contrast agent. This contrast agent will be injected into the arm and will help the doctors to read the MRI more effectively. If there is a lesion (abnormality) in the breast, the contrast agent will go to the lesion first and we will be able to see it better.
  The examination table will then move subject into the magnet, which is a long tube with a diameter of about 3 feet. Subject will be asked to lie in the magnet for about 15 minutes. During the periods when we are taking pictures, we will ask subject to be as still as possible.
  Groups: MRI Unknown Cancer Status Group

SUMMARY:
The purpose of this study is to test an innovative MRI breast cancer screening method in women with mammographically dense breasts as well as other women with moderately increased cancer risk. MRI, combined with other methods of risk assessment, has potential to significantly improve sensitivity to cancer in dense breasts and detect cancer in all cases at a much earlier stage, with far fewer interval cancers than mammography. Previous tests of MRI sensitivity show that this screening could significantly increase the likelihood of detecting invasive cancers resulting in decreased mortality from breast cancer.

Suspicious lesions will be defined by the clinical interpretation of the breast MRI images performed by the attending breast radiologists. Based on the radiologist determination that the MRI findings are suspicious (these findings include masses, non-mass enhancement and foci), suspicious lesions will be assigned a Bi-Rads code specifying whether additional work up or biopsy is necessary. These are Bi-Rads codes 0, 4 and 5. False positive diagnosis should be minimized as all attending physicians reading breast MRI at this institution are fellowship trained in breast imaging.

ELIGIBILITY:
Inclusion Criteria:

* Women that have had a mammographically and/or sonographically identified finding that will require image guided biopsy
* Women between ages 40-74 with dense breasts having a mammogram
* Women identified as having an average or intermediate risk of breast cancer (defined as 10- 20% lifetime risk based on a clinical risk model).

Exclusion Criteria:

* Women with metallic implants
* Women that are claustrophobic
* Women that have a fear of needles or contrast
* Women that have had an allergic reaction to contrast in the past
* Women that are pregnant
* Women who are demonstrated to be at risk for an allergic reaction or nephrogenic systemic fibrosis (NSF)

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who have had a mammographically and/or sonographically identified finding that will require image guided biopsy.
  Women between ages 40-74 with dense breasts having a mammogram
  Women who have been identified as having an average or intermediate risk of breast cancer (defined as 10-20% lifetime risk based on a clinical risk model)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
True Positive | 1 day
  The abbreviated scan successfully determines a cancer, confirmed by biopsy.

SECONDARY OUTCOMES:
True Negative | 1 day
  The abbreviated scan successfully determines no cancers are present, as confirmed with mammography or a standard MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Mitchell Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT04877912/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT04877912/ICF_001.pdf